CLINICAL TRIAL: NCT02329821
Title: Change of Lactate Concentration During Hartmann Solution Infusion for Hepatic Resection
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gaab Soo Kim, professor, Samsung Medical Center
Other Study IDs: 2014-09-159
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Hepatocellular Carcinoma; Liver Disease
Keywords: lactate; hartmann solution; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HCC group: patients with hepatocellular carcinoma
  Interventions: Other: hartmann solution
- donor group: patient for liver transplantation donation
  Interventions: Other: hartmann solution

INTERVENTIONS:
Other: hartmann solution — hartmann solution infusion in patients for hepatic resection

SUMMARY:
The investigators are trying to investigate metabolism of lactate sourced from IV Hartmann's solution in patients with hepatocellular carcinoma(HCC) compared with a control group(donation for liver transplantation) with normal liver function. Second purpose of this study is finding the predictive factor of changing metabolism of lactate sourced from IV Hartmann's solution in patients with HCC.

DETAILED DESCRIPTION:
The liver is important in acid-base physiology and electrolyte balance. It is important because it is a metabolically active organ which may be either a significant net producer or consumer of hydrogen ions.

Lactate is produced in the peripheral tissues such as the muscles, skin, brain, and red blood cells and it is metabolized predominantly in the liver and kidneys, first to pyruvate and secondly to glucose. In the healthy liver, there is a net-uptake of lactate caused by gluconeogenesis, and the liver exhibits a higher net lactate clearance than any other organ anticipated to be up to 70% of the whole body clearance. Lactic acidosis will result if this hepatic metabolism is not adequate.

Hartmann's solution, which contains 28 mmol/l of lactate and has a pH of 6.5, has been extensively used to maintain and replace intravascular volume in a variety of anesthetic procedures. Excessive use of saline has been observed to result in hyperchloraemic acidosis - which has been identified as a potential side effect of saline based solutions. It has been suggested that the use of balanced electrolyte solutions may avoid this effect.

A previous study concerned that normal saline, which does not contain lactate, might be detrimental to liver donors because of an association with hyperchloremic metabolic acidosis.

Metabolism of lactate sourced from IV Hartmann's solution also results in a net consumption of H+, but as this lactate was associated with Na+, the overall result is a net bicarbonate production. Effectively, metabolism of this lactate results in generation of an equivalent amount of bicarbonate. The investigators are evaluating about the metabolism of lactate sourced from IV Hartmann's solution in patients with HCC and donor for liver transplantation (control group).

All patients underwent multiple medical assessments before surgery, including routine laboratory tests (complete blood counts, standard liver and renal function tests, coagulation tests, and viral serology), and electrocardiography, chest X-ray, hepatobiliary imaging, percutaneous liver biopsy, and indocyanine green retention testing (ICG test). Hartmann solution(Hartmann, Choongwae pharmaceutical, Seoul, Korea) solution is composed of 130 mmol/l sodium,109 mmol/l chloride, 4 mmol/l potassium,1.5 mmol/l calcium, and 28 mmol/l lactate, and has a pH of 6.5.

Briefly, anesthesia was induced with thiopental sodium (5 mg/kg), and vecuronium(0.15 mg/kg). Endotracheal intubation was performed, and general anesthesia was maintained with sevoflurane (2-3 vol% in 50% air and oxygen). Throughout the surgery, the patients are monitored electrocardiography, pulse oximetry, capnography, esophageal temperature, invasive arterial pressure (via a radial artery catheter). Fluid administration(Hartmann solution) begin upon arrival in the operating room with 5ml/kg/hour rate. Acid-base status and lactate, electrolyte, and hemoglobin concentrations were assessed immediately and 2 hour after induction of anesthesia. The infusion rate of fluid is 5ml/kg/hour. The reasons of that rate are intravenous crystalloid administration has been restricted during hepatic dissection at the request of the surgeon and the investigators considered about the requirement of fluid loss. Mean arterial blood pressure >60mmHg and urine output >0.5 ml/kg/h were maintained during anesthesia. When mean arterial blood pressure was < 60 mmHg, the volume of fluid administered was increased initially and/or intravenous ephedrine (5-10 mg) was injected, as appropriate. If it cannot maintain the hemodynamic stability and need more fluid administration, the investigators manage other fluid administration or inotropics, and the case is withdrawn.

Duration of 2 hours, volumes of Hartmann solution and the result of arterial blood gas analysis (Acid-base status and lactate, electrolyte, and hemoglobin concentrations were assessed immediately and 2 hour after induction of anesthesia) is recorded.

The investigators compare the change of lactate level of patients with HCC and a control group( donation for liver transplantation) with normal liver function. After evaluating metabolism of exogenous lactate, the investigators are trying to find the predictive factor (among liver profile lab, MELD score, INR, functional liver volume, ICG test) of changing metabolism of lactate sourced from IV Hartmann's solution in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular carcinoma

Exclusion Criteria:

* patients with diabetic mellitus
* patients with electrolyte inbalance
* patients with renal failure

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hepatocelluar carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
changes of lactate level | at 2hour after induction
  hartmann solution is infused 5ml/kg/hr for 2 hour

SECONDARY OUTCOMES:
changes of acid-base status | at 2hour after induction
  hartmann solution is infused 5ml/kg/hr for 2 hour, changes of pH, base excess, bicarbonate level

CONTACTS AND LOCATIONS:
Overall Officials: Gaab Soo Kim, M.D, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea